CLINICAL TRIAL: NCT00687895
Title: Quality Malaria Case Management In Under- Fives In Primary Health Care (Phc) Institutions In Bagamoyo And Kibaha Districts Of Coastal Tanzania:a Multicomponent Controlled Intervention Study
Brief Title: Improved Clinical and Microscopy Diagnosis at Primary Health Care in Tanzania
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Muhimbili University of Health and Allied Sciences (Other)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Zull Premji, professor, Muhimbili University College of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: HF2003
Record Dates: First submitted 2008-05-28; First posted 2008-06-02 (Estimated); Last update posted 2008-06-02 (Estimated); Status verified 2008-05

CONDITIONS: Malaria
Keywords: malaria microscopy primary health care children
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): training in clinical algorithm plus microscopy
  Interventions: Procedure: Clinical algorithm and microscopy diagnosis of malaria
- 2 (Experimental): clinical algorithm
  Interventions: Procedure: Clinical algorithm and microscopy diagnosis of malaria
- 3 (No Intervention): Control

INTERVENTIONS:
Procedure: Clinical algorithm and microscopy diagnosis of malaria — Clinical alogarithm
  The content of the package included
  1. description of signs and symptoms of malaria disease
  2. history taking relevant to malaria and physical examination
  3. identification of danger signs and severe illness for referral
  4. appropriate treatment
  5. counseling patients on the use of drugs.
  Malaria microscopy. contents
  1. make thick blood smears from patients with fever and stain with Giemsa
  2. identify and count malaria parasites
  3. maintain the microscope and store blood slides.
  Arms: 1; 2

SUMMARY:
General objective: To improve the quality of fever case management in children in government health facilities in Tanzania Hypothesis:The training of health workers, as well as provision, training and use of microscopes for malaria diagnosis will improve the treatment of clinical episodes of fever in children while reducing the amount and costs of drugs

DETAILED DESCRIPTION:
PHC facilities were eligible for the study if they were rural government owned; accessible by road during rainy season; and within 3 hours by car from Muhimbili University College of Health Sciences (MUCHS), Dar es Salaam

All children attending the 16 PHC facilities under the study during daytime were enrolled if they fulfilled the following criteria:

1. below five years of age
2. fever (temperature≥37.5◦C) and/or reported history of fever in last 2 days
3. able to return to the facility on day 7 after treatment or any other day if symptoms were to worsen or recur
4. the mother/guardian or caretaker consented to participate.

Patients with severe disease and/or general danger signs requiring inpatient care according to the IMCI guidelines were admitted or referred to the health centers or the district hospitals

ELIGIBILITY:
Inclusion Criteria:

1. below five years of age
2. fever (temperature≥37.5◦C) and/or reported history of fever in last 2 days
3. able to return to the facility on day 7 after treatment or any other day if symptoms were to worsen or recur
4. the mother/guardian or caretaker consented to participate

Exclusion Criteria:

a) N/A

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3131 (Actual)
Dates: Start 2003-07; Primary Completion 2004-03 (Actual); Study Completion 2004-03 (Actual)

PRIMARY OUTCOMES:
the proportion of study children receiving prescriptions of antimalarial drugs in the respective arms | Day 0

SECONDARY OUTCOMES:
prescriptions of antibiotics, cost of drugs | Day 0
health outcome of the patients | Day 1-6, day 7

CONTACTS AND LOCATIONS:
Overall Officials: Anders Bjorkman, MD, Study Director — Karolinska Institutet
Locations (1):
- dispensaries/health centers in Kibaha and Bagamoyo, Coast, Coast Region, Tanzania

REFERENCES:
- [Background] Bates I, Bekoe V, Asamoa-Adu A. Improving the accuracy of malaria-related laboratory tests in Ghana. Malar J. 2004 Nov 1;3:38. doi: 10.1186/1475-2875-3-38. PMID 15516269
- [Derived] Ngasala B, Mubi M, Warsame M, Petzold MG, Massele AY, Gustafsson LL, Tomson G, Premji Z, Bjorkman A. Impact of training in clinical and microscopy diagnosis of childhood malaria on antimalarial drug prescription and health outcome at primary health care level in Tanzania: a randomized controlled trial. Malar J. 2008 Oct 2;7:199. doi: 10.1186/1475-2875-7-199. PMID 18831737